CLINICAL TRIAL: NCT06651619
Title: Efficacy of Education Versus Education Plus Prescribed Fluid Intake on Hydration Status in High School Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2406
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Dehydration
Keywords: hydration; hypohydration; adolescent; athlete; sports; exercise; behavior; education; high school
MeSH Terms: conditions — Dehydration; Motor Activity; Behavior | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No hydration education or fluid prescription. Pre-practice urine specific gravity (USG), pre- and post-practice body mass, thirst scale measures. Fluid intake during practice (whatever the team is drinking) .
- Hydration Education between Week 1 and Week 2 (Experimental): In-depth education session regarding the effects of dehydration, the performance benefits of proper hydration, and how to properly hydrate before, during, and after activity. Pre-practice urine specific gravity (USG), pre- and post-practice body mass, thirst scale measures. Fluid intake during practice (whatever the team is drinking).
  Interventions: Other: Hydration Education
- Hydration Education between Week 1 and Week 2 plus Prescribed Hydration Week 2 (Experimental): In-depth education session regarding the effects of dehydration, the performance benefits of proper hydration, and how to properly hydrate before, during, and after activity. Pre-practice urine specific gravity (USG), pre- and post-practice body mass, thirst scale measures. Provided a standard amount of bottled water to drink the evening prior (1 liter) and in the two hours before practice (20 oz). Fluid intake will be recorded in an intake log. Subjects will be permitted to eat or drink whatever they like in addition to the prescribed fluid. Fluid intake during practice (whatever the team is drinking).
  Interventions: Other: Water; Other: Hydration Education

INTERVENTIONS:
Other: Water — Prescribed amount of bottled water the evening prior and 2 hours prior to team practice
  Arms: Hydration Education between Week 1 and Week 2 plus Prescribed Hydration Week 2
Other: Hydration Education — 30-60 minutes
  Arms: Hydration Education between Week 1 and Week 2; Hydration Education between Week 1 and Week 2 plus Prescribed Hydration Week 2

SUMMARY:
Sports science testing by investigators at Gatorade Sports Science Institute has revealed that many athletes arrive at practice with a high urine specific gravity indicating they are hypohydrated. Though the data showed that most athletes don't lose more than 2% of their body weight in sweat during a training session, it is not known what the cumulative effects of living and training in a hot environment are over the course of a week. Previous research has indicated that prescribing fluid intake is more effective than education in improving drinking behavior during exercise. No studies to date have compared the impact of fluid intake prescription versus education in adolescent boys and girls playing outdoor and indoor sports.

Comparing sexes and training environment may provide more clarity around potential barriers and challenges to proper hydration for each environment.

DETAILED DESCRIPTION:
This study will implement a parallel design with 4 sports team groups: 1) Indoor girls, 2) Indoor boys, 3) Outdoor girls, and 4) Outdoor boys. Each group of 36 per groups will be randomized into 1 of 3 conditions: 1) control (no intervention), 2) hydration education intervention, 3) prescribed hydration and education intervention. Athletes will be observed for three practices per week for 2 weeks. Practices are separated by at least 48 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males between the ages of 13-19 years old
2. Non-smoker
3. Currently enrolled in the IMG sports program
4. Able to give verbal and written informed consent for participation as well as obtain parental consent if <18 years of age
5. Must be fluent in English reading, writing, and speaking
6. Parental permission

Exclusion Criteria:

1. Expulsion from school for any reason
2. Leaving the IMG sports program
3. Pregnant or planning to become pregnant
4. Illness or injury that impacts sport participation or fluid balance
5. Taking any medication that impacts fluid balance
6. Participation in a clinical trial within past 30 days
7. Participation in any PepsiCo trial within past 6 months
8. Any condition the study investigator believes would interfere with eligibility following the study protocol, effect the study results, or put the subject at undue risk

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
urine specific gravity (USG). | Pre-practice x 3 practices in Week 1 and 3 practices in Week 2
  Assessed using hand-held refractometer, units recorded to the nearest 0.001

SECONDARY OUTCOMES:
Body weight | Change from pre-practice to post-practice x 3 practices in Week 1 and 3 practices in Week 2
  Assessed using Tanita portable scale, units recorded to the nearest 0.01 kg
Fluid intake Week 2 (measured for Prescription Group only) | Intake from evening before through post-practice x 3 practices in Week 2
  Assessed using beverage weight scale. Units recorded to the nearest 1 ml
Thirst questionnaire | Change from pre-practice to post-practice x 3 practices in Week 1 and 3 practices in Week 2
  6 items (thirst, pleasure to drink now, mouth feel, taste, stomach fullness, stomach sickness) each anchored from not at all to very, each on a 100 mm scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Osterberg, PhD, RD, Principal Investigator — PepsiCo R&D Life Sciences, Sports Science
Locations (1):
- Gatorade Sports Science Institute (GSSI) at IMG Sports Academy, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No